CLINICAL TRIAL: NCT03354845
Title: Deprescribing of Symptomatic Medications in Patients Receiving Rehabilitative or Subacute Care
Brief Title: Deprescribing of Symptomatic Medications in Rehabilitative or Subacute Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bright Vision Hospital (Other)
Responsible Party: Principal Investigator, Charissa Ee, Pharmacist, Bright Vision Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016/2149
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Polypharmacy; Adverse Drug Reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: The study was conducted as an open trial with two parallel groups. A total of 200 patients were randomized to an intervention (deprescribing) or control (usual care) group in a 1:1 ratio. Randomization of patients was performed after recruitment by an independent administrator using GraphPad randomization sequence software ©2017. Doctors were free to make any changes to patients' medication regimens as they wished in both groups.
Who Masked: Participant
Masking Description: Group assignment was made known to the pharmacists and doctors involved in the deprescribing study intervention. However, patients were not aware of which group they had been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (usual care) group (No Intervention): In the control group, doctors maintained the usual practice of medication review, altering and discontinuing medications as necessary, without receiving deprescribing recommendations from pharmacists.
- Deprescribing intervention group (Other): The five-step patient-centred deprescribing process was utilized in the intervention group.
  Interventions: Other: Deprescribing intervention

INTERVENTIONS:
Other: Deprescribing intervention — Pharmacists assessed the appropriateness of target symptomatic medications and potential for discontinuation. After discussion with pharmacists and consideration of patients' and caregivers' preferences regarding discontinuation or dose reduction, doctors would deprescribe these symptomatic medications. Symptom recurrence, adverse drug withdrawal events (ADWEs), and the need for drug re-initiation or initiation of new symptomatic control medications after deprescribing were monitored and documented in the 1st, 2nd and 6th weeks.
  Other Names: Systematic deprescribing; Deprescribing algorithm; Five-step patient-centred deprescribing process
  Arms: Deprescribing intervention group

SUMMARY:
Deprescribing is a systematic method of withdrawing potentially inappropriate or unnecessary medications and is warranted in the elderly due to the high prevalence of polypharmacy. In particular, symptomatic control medications, such as acid suppressants, laxatives and painkillers, are frequently prescribed and continued, though such medications are rarely needed on a long-term basis.

Therefore, the study objectives were to determine the cost savings, effects and feasibility of implementing a systematic process of deprescribing medications for symptomatic management, namely, acid suppressants, laxatives, analgesics, and antiemetics.

DETAILED DESCRIPTION:
Deprescribing is a systematic process of identifying and withdrawing drugs, which are potentially or currently causing more harm than benefit to patients, based on each individual patient's condition, treatment goals and level of functioning. Deprescribing needs to be patient-centric with shared decision-making between patients or caregivers and the multidisciplinary care team. Five distinct steps of deprescribing have been elucidated, and they comprise: 1) performing a comprehensive patient medical/medication history; 2) considering the overall risk and appropriateness of drugs; 3) assessing possibility of and planning drug discontinuation; 4) initiating and documenting drug discontinuation; and 5) monitoring effects and providing patient support.

Deprescribing is necessary in elderly aged 65 years and above due to the higher prevalence of polypharmacy and unnecessary and inappropriate medication use, compared to younger age groups. In Singapore, statistics from an acute restructured hospital in 2013 showed that 50 percent or more of inpatients were discharged with at least five chronic medications.

The discontinuation of medications has been trialled in earlier studies without causing significant adverse effects or symptom recurrence. Positive outcomes demonstrated include enhanced cognition, improved health and reduced falls. However, it is necessary to investigate the effects and feasibility of deprescribing in the present local setting, where healthcare perceptions, and associations between medication discontinuation and patient clinical outcomes may be different from other studied populations.

Therefore, this randomized controlled intervention study was conducted in a community hospital in Singapore to determine the cost savings, effects and feasibility of implementing a systematic process of deprescribing medications for symptomatic management, namely, acid suppressants, laxatives, analgesics, and antiemetics.

ELIGIBILITY:
Inclusion Criteria:

* All patients, regardless of age, who were on at least one of the following target symptomatic control medications for deprescribing: acid suppressants/proton pump inhibitors (PPIs), laxatives, analgesics (paracetamol, nonsteroidal anti-inflammatory drugs (NSAIDs), codeine, tramadol) and antiemetics

Exclusion Criteria:

* Patients with terminal illness or cancer and patients with documented clinically significant dementia and had no accompanying caregiver

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Cost savings | 6 weeks
  Reduction in the cost of one month of medications

SECONDARY OUTCOMES:
Number of medications | 6 weeks
  Reduction in the total number of medications
Change in bowel movement following deprescribing | 6 weeks
  Adverse effect of constipation indicated by no bowel movement in the past two days (BNO ≥2/7)
Adverse consequences of deprescribing | 6 weeks
  Symptom recurrence, adverse drug withdrawal events (ADWEs), and the need for deprescribed medications to be restarted or initiation of new symptomatic control medications after deprescribing
Feasibility of implementation | 6 weeks
  Time required to complete the deprescribing process and the limitations and challenges encountered

CONTACTS AND LOCATIONS:
Overall Officials: Charissa Ee (Pharmacist), Principal Investigator — Bright Vision Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott IA, Hilmer SN, Reeve E, Potter K, Le Couteur D, Rigby D, Gnjidic D, Del Mar CB, Roughead EE, Page A, Jansen J, Martin JH. Reducing inappropriate polypharmacy: the process of deprescribing. JAMA Intern Med. 2015 May;175(5):827-34. doi: 10.1001/jamainternmed.2015.0324. PMID 25798731
- [Background] Reeve E, Shakib S, Hendrix I, Roberts MS, Wiese MD. Review of deprescribing processes and development of an evidence-based, patient-centred deprescribing process. Br J Clin Pharmacol. 2014 Oct;78(4):738-47. doi: 10.1111/bcp.12386. PMID 24661192
- [Result] Garfinkel D, Zur-Gil S, Ben-Israel J. The war against polypharmacy: a new cost-effective geriatric-palliative approach for improving drug therapy in disabled elderly people. Isr Med Assoc J. 2007 Jun;9(6):430-4. PMID 17642388
- [Result] Reeve E, Andrews JM, Wiese MD, Hendrix I, Roberts MS, Shakib S. Feasibility of a patient-centered deprescribing process to reduce inappropriate use of proton pump inhibitors. Ann Pharmacother. 2015 Jan;49(1):29-38. doi: 10.1177/1060028014558290. Epub 2014 Nov 10. PMID 25385826
- See also: National Health System. Deprescribing: a practical guide. May 2015 — http://www.derbyshiremedicinesmanagement.nhs.uk/assets/Clinical_Guidelines/clinical_guidelines_front_page/Deprescribing.pdf